CLINICAL TRIAL: NCT00515775
Title: Influence of a Inhaled Corticosteroid Therapy Versus Corticosteroid + LABA Therapy on the FeNO of Asthmatic Children
Status: Completed | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Dr. Christian Vogelberg, University Children's Hospital, Technical University Dresden
Other Study IDs: D5890L00015
Record Dates: First submitted 2007-08-13; First posted 2007-08-14 (Estimated); Last update posted 2009-02-13 (Estimated); Status verified 2008-10

CONDITIONS: Allergic Asthma

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective

SUMMARY:
The purpose of the study is to investigate, whether the FeNO concentration of asthmatic children is influenced differently by inhaled corticosteroid compared to inhaled corticosteroid + long acting beta agonist. The study hypothesis is that the FeNO concentration is more decreased in patients with a combination therapy compared to those with a corticosteroid mono therapy.

ELIGIBILITY:
Inclusion Criteria:

* allergic asthma since > 6 months equal or lower corticosteroid therapy before study entry FEV1>50%

Exclusion Criteria:

* severe asthma respiratory infection within the last 4 weeks smoking

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Allergic asthmatics
Sampling Method: Probability Sample
Enrollment: 27 (Estimated)
Dates: Start 2005-09; Primary Completion 2008-06 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Vogelberg, MD, Principal Investigator — University Children´s Hospital, Technical University of Dresden
Locations (1):
- University Children´s Hospital, Technical University of Dresden, Dresden, Germany